CLINICAL TRIAL: NCT00185302
Title: Phase II Study of MS-275, a Histone Deacetylase Inhibitor, Comparing 2 Dosage Schedules in Patients With Metastatic Melanoma
Brief Title: Safety and Efficacy Study of a New Chemotherapy Agent to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91410; 2004-002395-41 (EudraCT Number); 309100 (Other: Company ID)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Melanoma
Keywords: Non-resectable metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Histone Deacetylase Inhibitors; entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Histone Deacetylase Inhibitor, 3 mg (Experimental): Subjects received 3 mg MS-275 orally biweekly (Days 1 and 15 of a 4 week cycle) or until disease progression or unacceptable toxicity
  Interventions: Drug: Histone Deacetylase Inhibitor, MS-275 (BAY 86-5274, ZK 244894)
- Histone Deacetylase Inhibitor, 7 mg (Experimental): Subjects received 7 mg MS-275 orally weekly (Days 1, 8, and 15 of a 4 week cycle) until disease progression or unacceptable toxicity
  Interventions: Drug: Histone Deacetylase Inhibitor, MS-275 (BAY 86-5274, ZK 244894)

INTERVENTIONS:
Drug: Histone Deacetylase Inhibitor, MS-275 (BAY 86-5274, ZK 244894) — MS-275, 3 mg on Days 1 and 15 of a 4-week cycle
  Arms: Histone Deacetylase Inhibitor, 3 mg
Drug: Histone Deacetylase Inhibitor, MS-275 (BAY 86-5274, ZK 244894) — MS-275, 7 mg on Days 1, 8 and 15 of a 4-week cycle
  Arms: Histone Deacetylase Inhibitor, 7 mg

SUMMARY:
Primary objective: To evaluate the efficacy of two different dosing schedules of MS-275 in subjects with metastatic melanoma Secondary objectives: To evaluate the safety and to assess the pharmacokinetic profile of MS-275 in subjects with metastatic melanoma

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with Stage III or IV non-resectable nonuveal (cutaneous or mucosal) metastatic melanoma who had received at least one but no more than two previous systemic therapies (immunotherapy and/or chemotherapy) for metastatic disease and who had not responded to or who had progressed after their most recent therapy were eligible for enrollment
* Presence of at least one lesion fulfilling the minimum Response Evaluation Criteria in Solid Tumors (RECIST) size requirements for a target lesion - Use of highly effective birth control methods in females of child-bearing potential
* Able to undergo either contrast enhanced computed tomography (CT) scan or contrast enhanced magnetic resonance imaging (MRI) scan for tumor assessment
* Life expectancy greater than 3 months
* Adequate organ and bone marrow functions as defined below: absolute neutrophil count ≥ 1500 /µL, platelets ≥ 100,000 /µL, creatinine ≤ 1.5 × upper limit of normal (ULN) or measured creatinine clearance of ≥ 60 mL/min x 1.73 m2 body surface area, total bilirubin ≤ 1.5 times ULN, aspartate aminotransferase or serum glutamic oxalacetic transaminase/alanine aminotransferase or serum glutamic pyruvic transaminase∗ ≤ 2.5 times ULN
* Negative serum pregnancy test within 2 weeks prior to receiving the first dose of study drug in female subjects of childbearing potential. Agreement to use a highly effective method of birth control throughout the study period and 3 months thereafter for sexually active males and females of childbearing potentia

Exclusion Criteria:

* Active malignancy in the last five years
* Pregnancy, breast feeding
* HIV infection
* Brain metastasis
* Concomitant use of corticosteroids or valproic acid
* Uncontrolled intercurrent illness
* Diagnosis of uveal melanoma
* Eastern Cooperative Oncology Group performance status ≥ 2
* Ongoing effects from previous investigational drug studies or concomitant participation in other investigational drug studies
* Prior use of MS-275 or any other HDAC inhibitor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MS-275
* Anticancer therapy
* Active gastrointestinal conditions that might predispose for poor drug absorption
* Major surgery within 4 weeks prior to enrollment
* Hypophosphatemia < 2.5 mg/dL at screening, if not corrected in the screening period
* Medical, psychiatric or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-12; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Overall tumor response rate (the proportion of subjects with the best tumor response of PR or CR within the first 6 cycles of treatment) | Baseline, 8, 16, 24, 32 weeks (cycle 6)

SECONDARY OUTCOMES:
Time to tumor progression | Baseline, every 8 weeks until progression
Survival | At 6 months
Tumor response rate at each tumor assessment time point (CR/PR/SD/PD/not assessable) | At baseline and repeated every 2 cycles until tumor progression between Day 22 of even numbered cycles and Day 1 of subsequent odd numbered cycle and also at EOT and F-up visiit (90 days after the EOT and every 3 months until disease progression)
Time to death | Baseline, every 8 weeks until death
Number of participants with adverse events | Approximately 8-64 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/